CLINICAL TRIAL: NCT04410718
Title: Glycaemia and Cardiac Function in Patients With COVID-19
Acronym: GLYCOVID-19
Status: Completed | Type: Observational
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Andreas Andersen, Principal Investigator, Steno Diabetes Center Copenhagen
Other Study IDs: H-20024279
Record Dates: First submitted 2020-05-05; First posted 2020-06-01 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; COVID
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The intensive care unit cohort: Patients (with or without diabetes) with COVID-19 admitted to the intensive care unit
  Interventions: Other: Glycaemic levels
- The hospitalisation cohort: Patients with diabetes and COVID-19 admitted to the medical ward
  Interventions: Other: Glycaemic levels

INTERVENTIONS:
Other: Glycaemic levels — Glycaemic levels during admission for COVID-19

SUMMARY:
The study design is observational, exploratory study consisting of two cohorts of COVID-19 patients admitted to the ICU and the medical ward, respectively. The primary outcome focusing on the effect of plasma glucose levels on cardiac function will be evaluated by repeated assessment of cardiac function by echocardiography and measurement of plasma glucose. Furthermore, blood coagulability will be evaluated to determine the importance of diabetes status and plasma glucose changes for whole blood coagulability at time of admission to the ICU and progression in coagulability abnormalities. In the medical ward cohort, two assessments will be performed separated by no more than 12 hours. In the ICU cohort, three assessments will be performed separated by no more than 6 hours. Ideally, 60 patients with COVID-19 will be included in the ICU cohort with a 1:1 distribution between patient with and without diabetes. Ideally, 40 patients with diabetes will be included in the cohort of patients admitted to medical ward (hospitalisation cohort).

The primary hypothesis is that levels of plasma glucose have clinically significant impact on left ventricular systolic function in patients with COVID-19 admitted to the ICU. The secondary hypothesis is that the impact of plasma glucose on left ventricular systolic function is associated with glycaemic control prior to admission as measured by HbA1c.

ELIGIBILITY:
The ICU cohort - Inclusion criteria

* Informed and written consent
* Age ≥18 years
* Verified COVID-19
* Admission to the ICU within the last 24 hours
* Type 1 or type 2 diabetes prior to admission (the diabetes sub-group only)

The ICU cohort - Exclusion criteria

* Cardiac arrhythmia at time of inclusion (previously diagnosed paroxysmal atrial fibrillation will be allowed)
* Pacemaker rhythm
* Severe valve disease

The hospitalisation cohort - inclusion criteria

* Informed and written consent
* Age ≥18 years
* Verified COVID-19
* Admission to medical ward within the last 24 hours
* Type 1 or type 2 diabetes prior to admission

The hospitalisation cohort - Exclusion criteria

* Cardiac arrhythmia at time of inclusion (previously diagnosed paroxysmal atrial fibrillation will be allowed)
* Pacemaker rhythm
* Severe valve disease

Withdrawal criteria

- The participants may withdraw at will at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present study aims to evaluate the effect of glycaemia on cardiac function in patients with COVID-19 by examining cardiac function by echocardiography in two patient groups: 1) hospitalised COVID-19 patients with diabetes admitted to the medical ward 2) COVID-19 patients with or without diabetes admitted to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Plasma glucose levels and left ventricular ejection fraction | The study applies a mixed model for assessment of within-subject effects by repeated assessment in same individual. The time frame is from first assessment until last assessment (max. 24 hours).
  The within-subject effect of plasma glucose levels on left ventricular systolic function as measured by left ventricular ejection fraction (a pooled analysis of the hospitalisation cohort and ICU cohort)

SECONDARY OUTCOMES:
Key secondary outcome: HbA1c, plasma glucose levels and left ventricular systolic function | The study applies a mixed model for assessment of within-subject effects by repeated assessment in same individual. The time frame is from first assessment until last assessment (max. 24 hours).
  Difference in the within-subject effect of plasma glucose levels on left ventricular systolic function as measured by left ventricular ejection fraction between patients with chronic hyperglycaemia prior to admission (HbA1c >53 mmol/mol) and with normoglycaemia prior to admission (HbA1c ≤53 mmol/l) (ICU cohort only)
Plasma glucose levels and strain analysis | The study applies a mixed model for assessment of within-subject effects by repeated assessment in same individual. The time frame is from first assessment until last assessment (max. 24 hours).
  The within-subject effect of plasma glucose levels on left ventricular systolic function as measured by strain analysis (a pooled analysis of the hospitalisation cohort and ICU cohort)
Plasma glucose levels and mitral annular systolic velocity | The study applies a mixed model for assessment of within-subject effects by repeated assessment in same individual. The time frame is from first assessment until last assessment (max. 24 hours).
  The within-subject effect of plasma glucose levels on left ventricular systolic function as measured by mitral annular systolic velocity (a pooled analysis of the hospitalisation cohort and ICU cohort)
Plasma glucose levels and left ventricular ejection fraction (sub-group analysis) | The study applies a mixed model for assessment of within-subject effects by repeated assessment in same individual. The time frame is from first assessment until last assessment (max. 24 hours).
  Differences in the within-subject effect of plasma glucose levels on left ventricular systolic function as measured by left ventricular ejection fraction between the hospitalisation cohort, the ICU cohort with diabetes and the ICU cohort without diabetes, respectively
Plasma glucose levels and strain analysis (sub-group analysis) | The study applies a mixed model for assessment of within-subject effects by repeated assessment in same individual. The time frame is from first assessment until last assessment (max. 24 hours).
  Differences in the within-subject effect of plasma glucose levels on left ventricular systolic function as measured by strain analysis between the hospitalisation cohort, the ICU cohort with diabetes and the ICU cohort without diabetes, respectively
Plasma glucose levels and mitral annular systolic velocity (sub-group analysis) | The study applies a mixed model for assessment of within-subject effects by repeated assessment in same individual. The time frame is from first assessment until last assessment (max. 24 hours).
  Differences in the within-subject effect of plasma glucose levels on left ventricular systolic function as measured by mitral annular systolic velocity between the hospitalisation cohort, the ICU cohort with diabetes and the ICU cohort without diabetes, respectively
HbA1c, Plasma glucose levels and strain analysis | The study applies a mixed model for assessment of within-subject effects by repeated assessment in same individual. The time frame is from first assessment until last assessment (max. 24 hours).
  Difference in the within-subject effect of plasma glucose levels on left ventricular systolic function as measured by strain analysis between patients with chronic hyperglycaemia prior to admission (HbA1c >53 mmol/mol) and with normoglycaemia prior to admission (HbA1c ≤53 mmol/l) (ICU cohort only)
HbA1c, Plasma glucose levels and mitral annular systolic velocity | The study applies a mixed model for assessment of within-subject effects by repeated assessment in same individual. The time frame is from first assessment until last assessment (max. 24 hours).
  Difference in the within-subject effect of plasma glucose levels on left ventricular systolic function as measured by mitral annular systolic velocity between patients with chronic hyperglycaemia prior to admission (HbA1c >53 mmol/mol) and with normoglycaemia prior to admission (HbA1c ≤53 mmol/l) (ICU cohort only)
Diabetes status and whole blood coagulability and fibrinolysis | At time of admission to the ICU (max. 24 hours after admission to the ICU)
  Difference in whole blood coagulability and fibrinolysis as measured by TEG between patients with and without diabetes at time of admission to the ICU (ICU cohort only)
Diabetes status and change in whole blood coagulability and fibrinolysis during ICU stay | From first until last assessment during ICU stay (max. 24 hours).
  Difference in change in whole blood coagulability and fibrinolysis as measured by TEG between patients with and without diabetes treated at the ICU (ICU cohort only)
Prognostic value of TEG analysis | From time of admission and until four weeks after admission
  The prognostic value of cardiac function and TEG on the following patient outcomes 1) need for treatment in the ICU (hospitalisation cohort only) 2) need for respirator treatment (hospitalisation cohort only) 3) COVID-19 related death
Prognostic value of cardiac function | From time of admission and until four weeks after admission
  The prognostic value of cardiac function on the following patient outcomes 1) need for treatment in the ICU (hospitalisation cohort only) 2) need for respirator treatment (hospitalisation cohort only) 3) COVID-19 related death
Diabetes status and high-sensitivity troponins | At the time of admission to the ICU (max. 24 hours after admission to the ICU)
  Difference in cardiac damage as measured by high-sensitivity troponin (hs-troponin) between patients with and without diabetes admitted to the ICU (ICU cohort only)
Diabetes status and change high-sensitivity troponins | From first until last assessment during ICU stay (max. 24 hours)
  Difference in change in cardiac damage as measured by high-sensitivity troponin (hs-troponin) between patients with and without diabetes admitted to the ICU (ICU cohort only)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Herlev and Gentofte Hospital, Hellerup, Please Select
  - Hvidovre Hospital, Hvidovre, Please Select